CLINICAL TRIAL: NCT04914676
Title: Accelerated Dose Schedule of Cytarabine Consolidation Therapy for Patients With Acute Myeloid Leukemia (AML) in Complete Remission
Brief Title: Accelerated Dose Schedule of Cytarabine Consolidation Therapy for Older Patients With Acute Myeloid Leukemia (AML) in Complete Remission
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI decision to close study early due to limited data due to accrual goal not being met
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF-HEM-009; IRB202003214 (Other: University of Florida); OCR40160 (Other: University of Florida)
Record Dates: First submitted 2021-06-03; First posted 2021-06-04 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; high dose cytarabine; HiDAC; consolidation; chemotherapy schedule; bone marrow; elderly
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prospective HiDAC Treatment (HiDAC 123) (Experimental): Subject on this arm will be treated with HiDAC prospectively.
  Interventions: Drug: Cytarabine
- Historical HiDAC Treatment (HiDAC 135) (Other): Subjects on this arm will be historical controls who have previously received treatment with HiDAC.
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Drug: Cytarabine — Subjects on this arm will prospectively receive consolidation therapy with cytarabine. Subjects will be treated with 1000 mg/m2 cytarabine intravenously every 12 hours on Days 1-3 of each consolidation cycle. Subjects will receive up to four consolidation cycles.
  Other Names: Cytosar; cytosine arabinoside; Ara-C
  Arms: Prospective HiDAC Treatment (HiDAC 123)
Drug: Cytarabine — Subjects on this arm will have received consolidation therapy with cytarabine between 2/1/2017 and 2/1/2019. Subjects will have received 1000 mg/m2 cytarabine intravenously every 12 hours on days 1, 3, and 5 of each consolidation cycle and will have received up to 4 consolidation cycles.
  Other Names: Cytosar; cytosine arabinoside; Ara-C
  Arms: Historical HiDAC Treatment (HiDAC 135)

SUMMARY:
This phase 2, open label, non-randomized study will evaluate the safety of administering high dose cytarabine (HiDAC) consolidation therapy on days 1-3 of each cycle, as compared to standard administration on days 1, 3, and 5 of each cycle, in patients 61 years and older with de novo acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Both males and females ≥ 61 years of age
* A clinical diagnosis of de novo, non-M3 acute myeloid leukemia (AML) confirmed by greater than 20% blasts in peripheral blood or on diagnostic bone marrow biopsy who have completed intensive induction chemotherapy and are confirmed in complete remission #1 (defined by < 5% myeloblasts on recovery bone marrow biopsy, Absolute neutrophil count > 1000/uL and platelets > 100x103/uL) and able to receive HiDAC consolidation #1
* Patients on the prospective arm must be willing to have labs/clinic visits at UF Health Shands approximately every 48 hours +/- 24 hours after discharge from chemotherapy admission to be included. If prospective subjects cannot be followed at the UF site then telephone visits are allowed to follow for toxicity and transfusions. Records can be requested from subject's local physician office.
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures. For subjects on the historical arm, there will be a waiver of informed consent (as these patients may be deceased or not be available for retrospective consent).

Exclusion Criteria:

* Age < 61 years
* Patients unable to provide informed consent for prospective arm
* Secondary AML (documented history of antecedent hematological disorder, such as myelodysplastic syndrome or therapy-related AML) or chronic myeloid leukemia (CML) in blast crisis
* Patients receiving, received, or who will receive a FLT3 inhibitor
* Patients receiving, received, or who will receive an IDH1 or IDH2 inhibitor
* Serum creatinine greater than 2 mg/dL
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness
* For historical arm, subjects will be excluded if adequate data is not available in electronic medical record (e.g., if patient was followed by their local oncologist between chemotherapy cycles and labs/transfusions/clinic notes, etc. are not available)
* Karnofsky performance status of 40 or less at study entry

Ages: 61 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Hsu, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prospective HiDAC Treatment (HiDAC 123) | Historical HiDAC Treatment (HiDAC 135)
Started | 5 | 0 (No participants were enrolled on this arm because the study was terminated prior to any participants being enrolled on this arm.)
Completed | 2 | 0
Not Completed | 3 | 0
Not completed — Study termination | 3 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled on the historical arm because the study was terminated prior to any participants being enrolled on this arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective HiDAC Treatment (HiDAC 123) | Historical HiDAC Treatment (HiDAC 135) | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Full Range); unit: years] | 66.8 [61 to 73] |  | 66.8 [61 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  | 4
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 5 |  | 5
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 4 |  | 4
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Duration of Neutropenia
Description: Determine the duration of neutropenia in older patients with de novo AML after consolidation chemotherapy with HiDAC 123, as compared to historical controls treated with HiDAC 135.
Time Frame: 5 months
Population: Data were not collected for subjects on either arm. No subjects were enrolled on the historical control arm.
Arm/Group | Prospective HiDAC Treatment (HiDAC 123) | Historical HiDAC Treatment (HiDAC 135)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Duration of Thrombocytopenia
Description: Determine the duration of thrombocytopenia in older patients with de novo AML after consolidation chemotherapy with HiDAC 123, as compared to historical controls treated with HiDAC 135.
Time Frame: 5 months
Population: Data were not collected for subjects on either arm. No subjects were enrolled on the historical control arm.
Arm/Group | Prospective HiDAC Treatment (HiDAC 123) | Historical HiDAC Treatment (HiDAC 135)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Documented Infections
Description: Compare the incidence of documented infections (bloodstream infection, pneumonia, invasive fungal infection, Clostridium difficile infection, typhlitis, and febrile neutropenia) in patients receiving HiDAC 123 and HiDAC 135.
Time Frame: 5 months
Population: Data were not collected for subjects on either arm. No subjects were enrolled on the historical control arm.
Arm/Group | Prospective HiDAC Treatment (HiDAC 123) | Historical HiDAC Treatment (HiDAC 135)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Transfusions
Description: Compare the number of red blood cell and platelet transfusions per cycle in patients receiving HiDAC 123 and HiDAC 135.
Time Frame: 4 months
Population: Data were not collected for subjects on either arm. No subjects were enrolled on the historical control arm.
Arm/Group | Prospective HiDAC Treatment (HiDAC 123) | Historical HiDAC Treatment (HiDAC 135)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Readmission Rates and Length of Readmission Stay
Description: Compare the incidence of readmission and the length of readmission stay in patients receiving HiDAC 123 and HiDAC 135.
Time Frame: 5 months
Population: Data were not collected for subjects on either arm. No subjects were enrolled on the historical control arm.
Arm/Group | Prospective HiDAC Treatment (HiDAC 123) | Historical HiDAC Treatment (HiDAC 135)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Next Treatment
Description: Compare the time to next treatment (next chemotherapy cycle, transplant, etc.) in patients receiving HiDAC 123 and HiDAC 135.
Time Frame: 5 months
Population: Data were not collected for subjects on either arm. No subjects were enrolled on the historical control arm.
Arm/Group | Prospective HiDAC Treatment (HiDAC 123) | Historical HiDAC Treatment (HiDAC 135)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent until 28 days after the last dose of study treatment or the start of a new chemotherapy regimen (whichever came first). Adverse event data were collected for a maximum of 165 days.
Description: Adverse events were assessed by the principal investigator, the treating sub-investigator, and/or the study coordinator from the time of informed consent until 28 days after the last dose of study treatment or the start of a new chemotherapy regimen (whichever came first). Adverse events were assessed by physical examination, labs, and subject self-reports.
Arm/Group | Prospective HiDAC Treatment (HiDAC 123) | Historical HiDAC Treatment (HiDAC 135)
All-Cause Mortality (participants affected / at risk) | 2/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/5 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective HiDAC Treatment (HiDAC 123) (N=5) | Historical HiDAC Treatment (HiDAC 135) (N=0)
Altered mental status (Nervous system disorders) | 1 | NA
Anemia (Blood and lymphatic system disorders) | 1 | NA
Lung infection (Infections and infestations) | 1 | NA
Platelet count decreased (Investigations) | 1 | NA
Meningoencephalitis (Infections and infestations) | 1 | NA
Sepsis (Infections and infestations) | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prospective HiDAC Treatment (HiDAC 123) (N=5) | Historical HiDAC Treatment (HiDAC 135) (N=0)
Absolute neutrophil count decreased (Investigations) | 1 | NA
Alanine aminotransferase increased (Investigations) | 1 | NA
Altered mental status (Nervous system disorders) | 1 | NA
Anemia (Blood and lymphatic system disorders) | 5 | NA
Lymphocyte count decreased (Investigations) | 5 | NA
Neutrophil count decreased (Investigations) | 4 | NA
Platelet count decreased (Investigations) | 5 | NA
White blood cell decreased (Investigations) | 5 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT04914676/Prot_SAP_000.pdf